CLINICAL TRIAL: NCT05423158
Title: Virtual Care Strategies to Improve Participation in Cardiac Rehabilitation Among Veterans
Acronym: IMPACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Atlanta VA Medical Center (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); VA Ann Arbor Healthcare System (U.S. Federal Agency); Malcom Randall VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR 21-026
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Cardiac Rehabilitation; Telemedicine; Telerehabilitation; Veterans
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The investigators propose a randomized clinical trial evaluating the effects of HBCR alone (usual care) versus HBCR + d-Coaching. d-Coaching includes a private group for intervention participants with direct messaging on the Connecteam mobile app and engagement sessions via VA Video Connect.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- d-Coaching (Experimental): Will receive home-based cardiac rehabilitation (HBCR) with digital coaching (d-Coaching) intervention
  Interventions: Behavioral: d-Coaching
- Usual Care (No Intervention): Will receive home-based cardiac rehabilitation (HBCR) alone

INTERVENTIONS:
Behavioral: d-Coaching — MOVN mobile app: Each participant will be assigned a secure login account that does not include personal information for research only. Participants will be trained on how to access and use the MOVN private social network group.
  Annie text messaging: Participants will be registered in the Annie VA text messaging program to receive tailored, interactive "push" messages with a combination of 1 and 2-way tailored messages on goals, barriers, self-management, etc. (based on data collected in real-time from the Fitbit and barriers identified at baseline).
  Fitbit wearable device & mobile app: The intervention group will be instructed to use the Fitbit for step counts and maximizing the Fitbit mobile app/desktop platform to track all PA, sharing one's Fitbit profile with others (optional leaderboard), and use of all available features.
  Other Names: Digital Coaching
  Arms: d-Coaching

SUMMARY:
Home-based CR (HBCR) is an alternative to traditional CR programs that has comparable efficacy in improving morbidity/mortality and increases access to critical services. There is major potential to improve Veteran engagement in CR by combining digital coaching (d-Coaching) with existing VA-supported technologies. The investigator's theory-based intervention targets a critical component of successful CR engagement that is not available through traditional programs: virtual social support through a social network. In addition, the investigators propose to improve self-efficacy and self-regulation through interactive digital multi-media education, personalized feedback, and motivation so that Veterans can complete the prescribed HBCR program and maintain physical activity long-term. This RCT will evaluate the effects of HBCR alone (usual care) versus HBCR + d-Coaching, including a private group with direct messaging on the Connecteam mobile application and bimonthly engagement sessions via VA Video Connect. The investigators will randomly assign 150 Veterans from 2 HBCR programs to a 3-month intervention. The addition of d- Coaching to existing digital technologies will be operationalized by using a private social media group to provide social support, education, personalized feedback, and motivation.

The investigators aim to determine the effect of the d-Coaching intervention on: a) the number of completed HBCR sessions over 3 months, b) functional capacity, c) physical activity, c) psychosocial outcomes, d) clinical outcomes, and e) social cognitive factors of self-efficacy, self-regulation, and perceived social support over 6 months. The investigators will also evaluate the extent to which self-efficacy, self-regulation, and perceived social support mediate the effect of the intervention on function and physical activity.

DETAILED DESCRIPTION:
Underutilization of cardiac rehabilitation (CR). Cardiovascular disease (CVD) is the leading cause of mortality for adults in developed countries, including Veterans. Despite the guideline recommendations for cardiac rehabilitation (CR) for patients with qualifying cardiovascular conditions, participation rates have been dismal over the decades without significant improvement, both within VA and non-VA programs. Only 16.3% of Medicare patients and 10.3% of Veterans participated in center-based CR (CBCR) between 2007 and 2011 after hospitalization for MI, percutaneous coronary intervention, or coronary artery bypass graft surgery. Participation in CR is especially low for older adults (Medicare beneficiaries), Veterans, women, and individuals from underserved populations. Completion of CR programs is also a major problem as 24% and 50% of participants drop-out from CR programs. Barriers for CBCR participation and adherence include considerable travel burden, co-pay for non-VHA programs, time away from work, or being the primary caregiver for children or older adults. Home-based CR (HBCR) and hybrid CR programs (combination of CBCR and HBCR) are alternative approaches to promote exercise and provide education that have been traditionally provided in CBCR. HBCR programs have been studied in depth showing equivalency to CBCR without increased adverse events. However, although the provision of HBCR has alleviated some of the barriers related to CBCR participation, barriers to participation in HBCR include: lack of peer social support, safety concerns for patients at higher risk, lack of face-to-face monitoring and communication, and less patient accountability. While completion rates are marginally higher for HBCR programs than center-based programs, less than half (48%) of Veterans participating in the investigator's SFVAMC HBCR program completed at least nine sessions, well above the VA average of 13%.

Home-based CR in the VA system. Across the VA, only 28% of VAMCs (35/124) have a CBCR program, and low participation is a significant problem with only 8.4% of Veterans participating in at least one session of CBCR at a VA or non-VA contracted site. A growing number of alternative HBCR and hybrid programs now exist in the VA health system after a recent initiative by the Office of Rural health (ORH) to sponsor the expansion of 30 alternative programs nationally. In addition, there have been accelerated efforts by VA CBCR programs to improve access to CR services remotely (equivalent to HBCR) due to the limits on in-person care from the COVID-19 pandemic. VA program evaluations have shown Veterans preferred HBCR compared to CBCR, and Veterans hospitalized at a facility with a HBCR program were 3 to 4 times more likely to participate in HBCR compared to any CBCR program.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years of age
2. History of cardiovascular disease that qualified participant for CR (MI, percutaneous coronary intervention, coronary artery bypass grafting, heart failure, valve surgery)
3. Referral to participate in home-based Phase II CR.

Exclusion Criteria:

1. Participation in center-based Phase II CR.
2. Cognitive impairment (per Mini-Cog)
3. Lack of English proficiency/literacy (Digital coaching will be conducted in English. Participants will need to speak/read English to receive intervention.)
4. Unstable clinical conditions (e.g., unstable arrhythmias or heart block, active infection, uncontrolled hypertension, decompensated heart failure, unstable angina, etc.)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
HBCR sessions | 3 months
  Number of completed home-based cardiac rehabilitation sessions

SECONDARY OUTCOMES:
Physical activity | 3 months
  Rapid Assessment of Physical Activity
Functional capacity | 3 months
  Sit-to-Stand Test
Sedentary time | 3 months
  1-item International PA Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Linda Grace Park, PhD MS NP, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA; Joe R. Nocera, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No